CLINICAL TRIAL: NCT01811810
Title: Phase 2/3 Study of Dose-escalated External Beam Radiation Therapy
Brief Title: Proton Therapy for High Risk Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 22812
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
Keywords: Men under the age of 75 with histologically confirmed high risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Androgen Antagonists; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- xrt and long term ADT (Other): Radiation therapy (XRT) and long term androgen deprivation therapy
  Interventions: Radiation: Radiation therapy (XRT); Other: Androgen Deprivation Therapy (ADT)
- xrt, chemotherapy and short term ADT (Other): radiation therapy (XRT), chemotherapy and short term ADT
  Interventions: Radiation: Radiation therapy (XRT); Other: Androgen Deprivation Therapy (ADT); Other: Chemotherapy

INTERVENTIONS:
Radiation: Radiation therapy (XRT)
Other: Androgen Deprivation Therapy (ADT)
Other: Chemotherapy
  Arms: xrt, chemotherapy and short term ADT

SUMMARY:
The most common treatment for men with high risk prostate cancer is radiation therapy (XRT) followed by long term androgen deprivation therapy (ADT). Long-term AD is toxic, with substantial metabolic, physical, mental and sexual side-effects. In this study, the investigators propose a treatment strategy to optimize the control of high risk prostate cancer by using dose-escalated external beam radiation (proton therapy or IMRT) concurrent with docetaxel and adjuvant short-course AD. The investigators hypothesize that this approach will be superior to the current standard of care and obviate the need for long term AD. In this study, subjects will be randomized to either XRT with long term ADT or XRT and chemotherapy and short term ADT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma (within 365 days of randomization).
* High-risk for recurrence as determined by evidence of at least one of the following: Gleason Score 8-10 PSA 20 T stage T3
* Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material; Gleason score must be in the range 2-10. 6 cores are strongly recommended.
* Clinical stages T1a- T3 N0 M0 as staged by the treating investigator. (AJCC Criteria 7th Ed.-appendix III).
* PSA values 50 ng/ml within 90 days prior to randomization. Must be completed prior to biopsy or at least 21 days after prostate biopsy.
* Absolute Neutrophil Count (ANC) 1,800 cells/mm³ within 90 days prior to randomization.
* Platelets 100,000 cells/mm³ within 90 days prior to randomization.
* Hemoglobin 10 g/dl within 90 days prior to randomization. 3.1.9 ALT, AST, and total bilirubin within 1.5 X institutional upper normal limits within 90 days prior to randomization.
* ECOG status 0-1 (appendix II) documented within 90 days of randomization.
* Patient must sign study specific informed consent prior to randomization. Note: consent for legally authorized representative is not permitted.
* Completed all requirements listed in section 4.0 within the specified time frames.
* Able to start treatment within 56 days of randomization.
* At least 18 years old and less than or equal to 75 years of age.
* Men of child-producing potential must be willing to consent to use effective contraception while on treatment and for at least 3 months afterwards.
* Medical oncology consultation prior to randomization and medically approved for chemotherapy treatment per protocol.

Exclusion Criteria:

* Evidence of distant metastasis.
* Pelvic lymph nodes 1.5 cm in greatest dimension unless the enlarged lymph node is biopsied and negative.
* Prior prostate cancer surgery including but not limited to prostatectomy, hyperthermia and cryosurgery.
* Prior pelvic radiation for their prostate cancer.
* Prior androgen suppression.
* Severe, active co-morbidity, defined as follows:
* Active rectal diverticulitis, Crohns disease affecting the rectum or ulcerative colitis. (Non-active diverticulitis and Crohns disease not affecting the rectum are allowed).
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
* Myocardial infarction within the last 6 months.
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of randomization.
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
* Prior allergic reaction to the drugs involved in this protocol.
* Existing peripheral neuropathy grade 2.
* Prior systemic chemotherapy for prostate cancer.
* History of proximal urethral stricture requiring dilatation.
* Major medical, addictive or psychiatric illness which in the investigators opinion,will prevent the consent process, completion of the treatment and/or interfere with follow-up.
* Evidence of any other cancer within the past 5 years and 50% probability of a 5 year survival. (Prior or concurrent diagnosis of basal cell or non-invasive squamous cell cancer of the skin is allowed.)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03 (Estimated); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Christodouleas, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Guttilla A, Bortolus R, Giannarini G, Ghadjar P, Zattoni F, Gnech M, Palumbo V, Valent F, Garbeglio A, Zattoni F. Multimodal treatment for high-risk prostate cancer with high-dose intensity-modulated radiation therapy preceded or not by radical prostatectomy, concurrent intensified-dose docetaxel and long-term androgen deprivation therapy: results of a prospective phase II trial. Radiat Oncol. 2014 Jan 14;9:24. doi: 10.1186/1748-717X-9-24. PMID 24423462